CLINICAL TRIAL: NCT02199782
Title: Pilot Study of Cognitive Assessment in Welsh Speakers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Conor Martin (Other Government)
Collaborators: Betsi Cadwaladr University Health Board (Other Government)
Responsible Party: Sponsor-Investigator, Conor Martin, Dr Conor Martin, National Health Service, United Kingdom
Organization: National Health Service, United Kingdom (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BCUHB - PS - CAWS - 1
Record Dates: First submitted 2014-07-15; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Cognitive Impairment - e.g. Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Welsh (Active Comparator): Participants will complete the cognitive assessment in Welsh and in English these will be compared to assess whether first language Welsh speakers perform better in Welsh.
  Interventions: Other: Welsh language Cognitive Assessment
- English (Active Comparator): Participants will complete the cognitive assessment in Welsh and in English these will be compared to assess whether first language Welsh speakers perform better in Welsh.
  Interventions: Other: Welsh language Cognitive Assessment

INTERVENTIONS:
Other: Welsh language Cognitive Assessment — This intervention may intervene by displaying a more realisitic reflection of the patient's cognitive ability by assessing the patient in their first language

SUMMARY:
19% of Wales' population speaks Welsh. Under the Welsh Language Act 1993, every public body providing services to the public in Wales has to prepare a scheme setting out how it will provide those services in Welsh.

Diagnosing dementia requires a comprehensive assessment, an essential component of which is a cognitive assessment tool, which takes the form of a questionnaire. In clinical practice, this is currently only available through the medium of English.

The investigators objective is to measure the difference between Cognitive Assessment scores (using the Montreal cognitive assessment (MoCA)), when done in English and Welsh, in those who are cognitively impaired and whose first language is Welsh. The investigators predict that there will be a significant difference in scores in favour of the Welsh-medium tests, thus proving that the current mode of administering the test is prejudiced against patients whose first language is Welsh.

If the investigators predictions are correct, then the investigators would seek to introduce a validated Welsh-language cognitive assessment tool to the domain of the Welsh NHS.

ELIGIBILITY:
Inclusion Criteria:

* Welsh Speakers - self-identify as first-language Welsh
* Diagnosis of Dementia - recorded in patient's case notes

Exclusion Criteria:

* Refusal
* Intercurrent illness
* Blind/any other disability which may prevent participant from fully completing Cognitive Assessment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-08 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Difference in Cognitive Assessment Score between Welsh and English | at 0 and 48 hrs

SECONDARY OUTCOMES:
To measure the differences between participants' scores in Welsh and English and compare between different types of Dementia | 0 and 48hrs
  We will records each participant's type of cognitive decline - e.g. Alzheimer's, Vascular, Frontal, Lewy Body, etc, and compare the differences in scores - to see whether different types of dementia will perform significantly worse or better in their first and second languages (Welsh and English).

CONTACTS AND LOCATIONS:
Overall Officials: Sion Jones, MBBCh, Principal Investigator — BCUHB NHS
Locations (1):
- Ysbyty Glan Clwyd, Bodelwyddan, Denbighshire, United Kingdom

REFERENCES:
- [Background] Cummings JL, Benson F, Hill MA, Read S. Aphasia in dementia of the Alzheimer type. Neurology. 1985 Mar;35(3):394-7. doi: 10.1212/wnl.35.3.394. PMID 3974897
- [Background] Mendez MF, Perryman KM, Ponton MO, Cummings JL. Bilingualism and dementia. J Neuropsychiatry Clin Neurosci. 1999 Summer;11(3):411-2. doi: 10.1176/jnp.11.3.411. No abstract available. PMID 10440021